CLINICAL TRIAL: NCT06207526
Title: Delusion Ideation in the Context of Everyday Life: a Novel Smartphone-supported Psychological Therapy Approach (DICE)
Brief Title: Delusion Ideation in the Context of Everyday Life
Acronym: DICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutscher Akademischer Austausch Dienst (Other); Swinburne University of Technology (Other)
Responsible Party: Principal Investigator, Kerem Böge, PD Dr. Dr., Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DICE2023
Record Dates: First submitted 2023-12-19; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Psychotic Disorder
Keywords: psychotic disorders; psychotherapy; EMA; EMI; delusions
MeSH Terms: conditions — Psychotic Disorders; Delusions

STUDY DESIGN:
Intervention Model Description: A single-arm-feasibility-design is used. All participants will receive the intervention immediately after the baseline assessment (T0). All participants are allowed to continue standard scheduled treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blended face-to-face and smartphone intervention for delusional thoughts and experiences (Experimental): The blended face-to-face and smartphone intervention is implemented as a four-session intervention that is primarily based on an intervention from Bell et al. (2018/2020) which focused on hallucinations and is now being tailored to delusions. The intervention itself builds on the "Coping Strategy Enhancement" - program by Tarrier and colleagues (CSE; (Tarrier et al., 1990) by systematically build upon already applied coping strategies and therefore improve coping with psychotic symptoms. Participants receive four therapy sessions in person, while the app is used to collect data between sessions to be used in therapy and to record and train coping strategies between sessions.
  All participants are allowed to continue parallel implemented standard scheduled treatment.
  Interventions: Behavioral: Blended face-to-face and smartphone intervention

INTERVENTIONS:
Behavioral: Blended face-to-face and smartphone intervention — The intervention comprises two phases: an initial stage involves baseline assessment, in-depth app training, psychoeducation, and EMA monitoring for functional analysis. The subsequent phase focuses on identifying and implementing individual coping strategies, forming the basis for daily personalized EMI reminders. Over six days, participants receive ten daily surveys to gauge fluctuations in paranoia and delusional ideation. EMA-derived feedback, considering antecedents and coping responses, shapes a personalized EMI. Four sessions with a psychologist involve discussing app feedback, emphasizing functional analysis, coding coping strategies into the app, assessing utility, and adapting as needed. Post-session two, five coping reminders and an eight-item evening survey are sent daily for two blocks of ten days to monitor delusional ideations and coping strategy effectiveness.

SUMMARY:
The project aims to investigate the feasibility and acceptability of a blended face-to-face and smartphone intervention for distressing thoughts and experiences in people with schizophrenia spectrum disorders. A secondary aim is to assess the outcomes of the intervention at baseline (T0) and post-intervention (T1) (single-arm feasibility design). The study design is primarily based on Bell et al.'s (2018, 2020) blended face-to-face and smartphone intervention for hallucinations. The participants receive four face-to-face therapy sessions, using a smartphone between sessions employing elements of Ecological Momentary Assessment (EMA) and Intervention (EMI).

DETAILED DESCRIPTION:
The investigators will identify eligible participants at different outpatient departments, suitable support groups, and online platforms. An eligibility screening conducted in person or by telephone to ensure the inclusion criteria and to introduce the study is held by the study assistant. All participants must sign an informed consent after written and verbal study clarification. Participants will carry out self-reported measurements at baseline (T0) and after the intervention phase of 4-6 weeks (T1). The group of participants receives four therapy sessions, using a smartphone between sessions.

The intervention begins with a session of psychoeducation, assessment and training, followed by a week of EMA monitoring using the participant's own smartphone or one provided by the research team. In the second session, EMA data will be discussed between therapist and participants to identify patterns in experiences, including effective and ineffective coping strategies. In the weeks between the remaining sessions, participants are reminded of these strategies via the app using EMI.

The data management plan includes standard procedures for data-handling such as using anonymized identification codes for patient data. Besides, the participants have the right to access their data, and the right to claim an annihilation. The data is being saved in an online database, only allowing researchers involved in the study to access the data.

ELIGIBILITY:
Inclusion Criteria:

1. be between 18 and 65 years old
2. fulfill the diagnostic criteria for schizophrenia as determined by the Mini-International Neuropsychiatric Interview (M.I.N.I.) (Sheehan et al., 1998)
3. suffer from residual delusions and significant self-reported distress as assessed by the PSYRATS Delusions (Haddock et al., 1999), Green Paranoid Thoughts, and Subjective Experiences of Psychosis Scales (Freeman et al., 2021).
4. sufficient knowledge of German
5. have not undergone a recent (<6 weeks) or planned change in antipsychotic and other psychopharmacological medication
6. know how to use a smartphone or be willing to learn how to use it
7. Time availability to attend 4 therapy appointments with two additional rating appointments

   Exclusion Criteria:
8. Severe visual impairment
9. Acute suicidal tendencies
10. Excessive delusional symptoms (Reference: 25+; Persecution: 28+ in the Green Paranoid Thoughts and Subjective Experiences of Psychosis Scales (Freeman et al., 2021)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of the intervention | Post-Intervention (after completion of 4 face-to-face psychotherapy sessions; 4-6 weeks from baseline)
  Feasibility will be indexed by completion rates of the EMA questionnaires (minimum threshold of >33% of completed EMA questionnaires), by whether participants use the application between sessions (>80% of clients) and whether the target level of ecological momentary assessment data for analysis is recorded (>80% of clients).
Acceptability of the intervention | Post-intervention (after completion of 4 face-to-face psychotherapy sessions; 4-6 weeks from baseline)
  Acceptability will be assessed by using the Client Satisfaction Questionnaire (Attkisson & Zwick, 1982) and a series of open-ended questions about elements of the intervention, in addition to the rate of intervention completion (>80% complete all sessions).
Side effects | Post-intervention (after completion of 4 face-to-face psychotherapy sessions; 4-6 weeks from baseline)
  Negative effects will be recorded by using the Negative Incidents and Effects Questionnaire (Rozental et al., 2019).

SECONDARY OUTCOMES:
Objective intensity of delusions | At baseline and post-intervention (after completion of 4 face-to-face psychotherapy sessions; 4-6 weeks from baseline)
  The psychotic symptom rating scales, PSYRATS (Haddock et al., 1999), measures the severity of different dimensions of auditory hallucinations and delusions, designed as semi-structured interviews. We will be using the delusions scale
Subjective intensity of delusions | At baseline and post-intervention (after completion of 4 face-to-face psychotherapy sessions; 4-6 weeks from baseline)
  The Green Paranoid Thought Scale in its revised form, R-GTPS (Freeman et al., 2021), will be used to record the subjective intensity of delusions. The measuring instrument consists of two separate subscales, with eight items assessing ideas of reference and ten items assessing ideas of persecution.
Psychological distress | At baseline and post-intervention (after completion of 4 face-to-face psychotherapy sessions; 4-6 weeks from baseline)
  The Subjective Experiences of Psychosis Scale, SEPS (Haddock et al., 2011), will be used to assess the psychological distress associated with experiencing delusions, as it is a measurement to assess an index of psychosis-related impact. The SEPS is a 41 item self-report scale assessing experiences of psychosis in terms of three subscales.
Stress, anxiety and depression | At baseline and post-intervention (after completion of 4 face-to-face psychotherapy sessions; 4-6 weeks from baseline)
  The Depression Anxiety Stress Scale (Nilges & Essau, 2015) will be used to analyse symptoms of stress, anxiety and depression.
self-assessed recovery | Post-intervention (after completion of 4 face-to-face psychotherapy sessions; 4-6 weeks from baseline)
  The Questionnaire about the Process of Recovery (Neil et al., 2009) will be used as a measure of self-assessed recovery of mental health.
Delusional ideation | At baseline, during EMA and post-intervention (after completion of 4 face-to-face psychotherapy sessions; 4-6 weeks from baseline)
  The 21-item Peters et al. (2004) Delusions Inventory (PDI) is being used to measure the delusional ideation. The PDI incorporates the multidimensionality of delusions by including measures of distress, preoccupation, and conviction. Participants have to rate their predominant pdi-item troughout the EMA.
Adverse events | Post-intervention (after completion of 4 face-to-face psychotherapy sessions; 4-6 weeks from baseline)
  The Negative Incidents and Effects Questionnaire (NIEQ) (Rozental et al., 2019) will be used to register adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No